CLINICAL TRIAL: NCT05633953
Title: A Retrospective Observational Study to Evaluate the Safety and Effectiveness of Osilodrostat for the Treatment of Non-Cushing's Disease Cushing's Syndrome (LINC7)
Brief Title: Osilodrostat for the Treatment of Non-Cushing's Disease Cushing's Syndrome
Acronym: LINC7
Status: Completed | Type: Observational
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Other Study IDs: LCI699-RECAG-NI-0596
Record Dates: First submitted 2022-11-16; First posted 2022-12-01 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Cushing's Syndrome
Keywords: Endogenous Cushing's Syndrome; Cushing's Syndrome; Osilodrostat
MeSH Terms: conditions — Cushing Syndrome | interventions — Osilodrostat

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Osilodrostat — oral administration

SUMMARY:
This is a multi-centre, observational, non-comparative, retrospective cohort study designed to evaluate the long-term safety and effectiveness of osilodrostat in non-CD CS patients. Patients treated with oral osilodrostat regardless of the duration of their treatment will be followed retrospectively for up to 36 months after initiating osilodrostat.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥18 years old with diagnosis of CS, except for CD (i.e., an aetiology of adrenal adenoma, adrenocortical carcinoma, adrenal hyperplasia, or ectopic adrenocorticotropic hormone secretion). Patients should have a contemporaneously documented diagnosis of CS as per effective guidelines.
2. Patients treated with osilodrostat between April 2019 and study start date as part of ATU programme or commercialisation.

Exclusion Criteria:

1. Patients who participated in a clinical trial anytime during the study period.
2. Patients with Pseudo-Cushing's syndrome, cyclic CS, or iatrogenic CS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with non-CD CS. Patients meeting eligibility criteria will be retrospectively identified and included in the study by site investigators based on a review of medical records at site. Site policies and local regulations regarding patient consent (NOL) will be followed. All eligible patients identified at a site between April 2019 and study start date and consenting to be part of the study will be included.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario M MALDONADO, MD, Study Director — RECORDATI GROUP
Locations (1):
- Hôpital Haut-Lévèque, Pessac, France

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Osilodrostat: Patients treated with oral osilodrostat regardless of the duration of their treatment or dosage followed retrospectively for up to 36 months after initiating osilodrostat. Followup of each patient was variable and based on the clinical judgement od the physicians
Period: Overall Study
Arm/Group | Osilodrostat
Started | 103 (1 screening failure)
Completed | 43
Not Completed | 60
Not completed — Adverse Event | 7
Not completed — Death | 30
Not completed — Lost to Follow-up | 1
Not completed — Osilodrostat discontinued | 4
Not completed — Physician Decision | 1
Not completed — Planned surgery related to Cushing Syndrome (CS) | 15
Not completed — Progressive disease | 2

BASELINE CHARACTERISTICS:
Groups:
- Osilodrostat: Patients treated with oral osilodrostat regardless of the duration of their treatment followed retrospectively for up to 36 months after initiating osilodrostat. Followup of each patient was variable and based on the clinical judgement od the physicians
Arm/Group | Osilodrostat
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (15.52)
Age, Customized [Count of Participants; unit: Participants]
  ≤ 65 years | 58
  ≥ 65 years | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 103
Height [Mean (Standard Deviation); unit: cm] — Population: Unable to collect for some patients
  cm
    number analyzed (Participants) | 99
    (all) | 166.7 (10.57)
Weight [Mean (Standard Deviation); unit: kg] — Population: Unable to collect data for some partecipants
  kg
    number analyzed (Participants) | 88
    (all) | 76.55 (22.295)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Unable to collect data from some partecipants
  kg/m^2
    number analyzed (Participants) | 86
    (all) | 27.77 (6.937)
Duration since CS diagnosis [Mean (Standard Deviation); unit: Months] | 14.27 (38.619)
CS causation [Count of Participants; unit: Participants]
  Adrenal Adenoma | 17
  Adrenocortical carcinoma | 19
  Adrenal hyperplasia | 14
  Ectopic ACTH secretion | 53

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Osilodrostat
Description: Number and proportion of patients with Mean Urinary Free Cortisol (mUFC) ≤ upper limit of normal (ULN)
Time Frame: at week 12
Population: Patients demonstrating a complete mUFC response at Week 12 with non-missing values
Measure: Count of Participants; unit: Participants
Groups:
- Osilodrostat_ITT: Patients treated with oral osilodrostat regardless of the duration of their treatment followed retrospectively for up to 36 months after initiating osilodrostat.
  Intent-to-treat (ITT) Population: All enrolled patients who had met all inclusion criteria and none of the exclusion criteria and received osilodrostat treatment for non-CD CS, with a potential follow-up of at least 12 weeks.
Arm/Group | Osilodrostat_ITT
Number analyzed (Participants) | 45
Participants | 23

2. Secondary Outcome: Long-term Effects of Osilodrostat on Mean Urinary Free Cortisol (mUFC)
Description: Proportion of patients with Mean Urinary Free Cortisol (mUFC) ≤ upper limit of normal (ULN) by visit until the earlier of loss to follow-up, treatment discontinuation, death and up to 36 months of retrospective follow-up.
Time Frame: at weeks 18, 24, 36, 48, 60, and 72
Population: Of all the patients, only the ones with non missing data at each visit were considered to analyse the variation on mUFC
Measure: Count of Participants; unit: Participants
Arm/Group | Osilodrostat
Number analyzed (Participants) | 21
Participants
  week 18: number analyzed (Participants) | 13
  week 18 | 7
  week 24 | 12
  week 36: number analyzed (Participants) | 10
  week 36 | 6
  week 48: number analyzed (Participants) | 7
  week 48 | 6
  week 60: number analyzed (Participants) | 9
  week 60 | 6
  week 72: number analyzed (Participants) | 7
  week 72 | 6

3. Secondary Outcome: Long Term Effects of Osilodrostat on Morning Serum Cortisol
Description: Proportion of patients with normal measures of morning serum cortisol [≤ upper normal limit (ULN)] by visit until the earlier of loss to follow-up, treatment discontinuation, death and up to 36 months of retrospective follow-up.
Time Frame: At baseline and Weeks 4, 8, 12, 18, 24, 36, 48, 60 and 72
Population: The analysis was done only on patients with no-missing data at each visit
Measure: Count of Participants; unit: Participants
Groups:
- Osilodrostat_ITT: Patients treated with oral osilodrostat regardless of the duration of their treatment followed retrospectively for up to 36 months after initiating osilodrostat.
Arm/Group | Osilodrostat_ITT
Number analyzed (Participants) | 56
Participants
  Baseline | 18
  week 4: number analyzed (Participants) | 44
  week 4 | 19
  week 8: number analyzed (Participants) | 12
  week 8 | 6
  week 12: number analyzed (Participants) | 42
  week 12 | 22
  week 18: number analyzed (Participants) | 20
  week 18 | 10
  week 24: number analyzed (Participants) | 24
  week 24 | 16
  week 36: number analyzed (Participants) | 16
  week 36 | 8
  week 48: number analyzed (Participants) | 11
  week 48 | 9
  week 60: number analyzed (Participants) | 14
  week 60 | 9
  week 72: number analyzed (Participants) | 9
  week 72 | 6

4. Secondary Outcome: Long-term Effects of Osilodrostat on Composite Cortisol Measure
Description: Proportion of patients with normal response of composite cortisol (salivary cortisol, urinary cortisol and morning serum cortisol) [≤ upper normal limit (ULN)] by visit until the earlier of loss to follow-up, treatment discontinuation, death and up to 36 months of retrospective follow-up.
Time Frame: At baseline and Weeks 4, 8, 12, 18, 24, 36, 48, 60 and 72
Population: Only the subjects with no-missing data at each visit were considered in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Osilodrostat_ITT
Number analyzed (Participants) | 68
Participants
  Baseline | 30
  week 4: number analyzed (Participants) | 54
  week 4 | 30
  week 8: number analyzed (Participants) | 17
  week 8 | 11
  week 12: number analyzed (Participants) | 55
  week 12 | 35
  week 18: number analyzed (Participants) | 24
  week 18 | 16
  week 24: number analyzed (Participants) | 30
  week 24 | 23
  week 36: number analyzed (Participants) | 20
  week 36 | 13
  week 48: number analyzed (Participants) | 12
  week 48 | 10
  week 60: number analyzed (Participants) | 16
  week 60 | 13
  week 72: number analyzed (Participants) | 9
  week 72 | 8

ADVERSE EVENTS:
Time Frame: For 36 months (study period) and for at least 12 weeks of retrospective follow-up (follow-up for each patient was variable, and based on the clinical judgement of the physicians at the investigative sites).
Arm/Group | Osilodrostat
All-Cause Mortality (participants affected / at risk) | 30/103
Serious Adverse Events (participants affected / at risk) | 52/103
Other Adverse Events (participants affected / at risk) | 87/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Osilodrostat (N=103)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adrenal insufficiency (Endocrine disorders) | 10
General physical health deterioration (General disorders) | 5
Death (General disorders) | 3
Multi organ dynsfunction syndrome (General disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 2
Presyncope (Nervous system disorders) | 3
Epilepsy (Nervous system disorders) | 2
Cardiac failure acute (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 2
COVID-19 (Infections and infestations) | 2
Acute kidney injury (Renal and urinary disorders) | 6
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Vascular disorders (Vascular disorders) | 4
Anemia (Blood and lymphatic system disorders) | 2
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1
Hepatobiliary disorders (Hepatobiliary disorders) | 1
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Osilodrostat (N=103)
Asthenia (General disorders) | 14
Oedema peripheral (General disorders) | 6
Adrenal insufficiency (Endocrine disorders) | 29
Diarrhoea (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 12
Abdominal pain (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 18
Acute kidney injury (Renal and urinary disorders) | 8
Hypertension (Vascular disorders) | 6
Anaemia (Blood and lymphatic system disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT05633953/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT05633953/SAP_001.pdf